CLINICAL TRIAL: NCT05778409
Title: To Study the Effects of Cordyceps Cicadae on Vision Care
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hui Wen Lin, Clinical Professor, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRREC-111-087
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cordyceps Cicadae extract group (Experimental): 500 mg/ day for 1 month
  Interventions: Biological: Cordyceps cicadae extract

INTERVENTIONS:
Biological: Cordyceps cicadae extract — 500mg/ day for one month

SUMMARY:
Cordyceps cicadae is a traditional Asian herbal medicine with a variety of bioactive substances and curative effects similar to Cordyceps Cicadae, and it has been reported that anti-dry eye and eye protection ingredients can be extracted. With the advancement of civilization, the number of patients with high myopia is increasing year by year and suffers from complications of dry eye or other eye diseases. In this study, the subjects were provided with cicadae extract or placebo in a double-blind manner, tracked the degree of visual fatigue by regular questionnaires, and measured for visual acuity, axial length and diopter. The purpose of this study is to investigate the effect of cicadae extract on visual acuity and visual fatigue, and to evaluate its potential as a health food ingredient.

DETAILED DESCRIPTION:
1. Visual acuity measurement: Snellen's Chart was used to measure visual acuity.
2. Refractive examination: Measure binocular refraction with Open Field computer refractor (Shin-Nippon Nvision K5001 Wide View).
3. Measuring the axial length of the eye: Use the multifunctional optical eyeball length measuring instrument (Lenstar) to measure the distance from the instrument to the optical paths such as the cornea, lens, and retina, and then convert to the axial length of the eye.
4. Corneal radian measurement: Use a keratometer (Bausch & Lomb Keratometer) to measure the corneal radian and curvature, and estimate the degree of corneal astigmatism.
5. Visual fatigue questionnaire survey: A visual fatigue scale questionnaire was designed using Ocular Surface Disease Index (OSDI) and Computer Vision Syndrome (CVS).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20 or over
2. Willing to participate in this study and sign the subject's consent form
3. Myopia less than 700 degrees

Exclusion Criteria:

1. Have consumed related eye care products in past 3 months
2. Those who have eye infection in the past 3 months
3. People who have been diagnosed with any eye diseases in past 3 months
4. Those who are allergic to cicadae

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Eye fatigue questionnaire | one month
  1. Eye fatigue were evaluated according to The Ocular Surface Disease Index (OSDI) introduced in 1997 by the Outcomes Research Group (Allergan Inc., Irvine, CA).
  2. Content including: (1) Eye swelling, (2) Eye soreness, (3) Photophobia, (4) Blurred vision, (5) Dry eye, (6) Foreign body sensation, (7) Tearing, (8) General discomfort related to eye fatigue.
  3. Scores are expressed on a scale of 0-3. 0 = No symptoms , 1 = Occasionally (≤1 time/day), 2 = Sometimes (1-3 times/day), 3 = Frequently (>3 times/day), a low score means less visual fatigue and better eye quality.
Best vision test | one month
  1. Visual acuity was tested with the Snellen Eye Test Chart and recorded with the score proposed by Snellen.
  2. Subjects were asked to stand 20 feet away to observe the snellen E-chart and record the smallest visual mark.
  3. Recording method: 20/20 (1.0) is defined as normal vision, lower than this score indicates that the subject has ametropia, and higher than this indicates that the subject's vision is higher than the general standard

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Wen Lin, Ph.D, Principal Investigator — Asia University
Locations (1):
- Asia university, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No